CLINICAL TRIAL: NCT01251952
Title: Phase I Dose Escalation Trial of Denileukin Diftitox (Ontak) Post Autologous Transplantation.
Brief Title: Dose Escalation Trial of Denileukin Diftitox (Ontak) Post Autologous Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug unavailable
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WSU 2010-039
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Denileukin Diftitox (Ontak) (Experimental): Denileukin Diftitox (Ontak) administered Post Autologous Transplantation.
  Interventions: Drug: Denileukin Diftitox (Ontak)

INTERVENTIONS:
Drug: Denileukin Diftitox (Ontak) — After receiving their stem cell transplant on Day 0, participants will receive study agent via a 30 minute infusion. Participants will also receive a 30 minute infusion of study agent on Day 21.
  Follow-up visits for clinical assessment, blood draws for routine clinical laboratory studies and for immuno-correlative studies will also take place on days 42, 90, 180 and 360.
  Other Names: Ontak®

SUMMARY:
The primary goal of this study is to determine the feasibility and safety of giving two doses of denileukin diftitox (DD) at days 0 and 21 post autologous stem cell transplantation in a dose escalation fashion. Secondary goals include evaluating the the effect of DD on the number and percentage of T-regs in the peripheral blood post transplant at each dose level, the effect of DD on T cell (CD4/CD8) reconstitution post transplant at each dose level and determining the time to engraftment: absolute neutrophil count (>0.5 x 10^9/L for 3 consecutive days), and platelet (>20X 10^9/L for 3 consecutive days).

The hypothesis for the study is based on the ability of DD to deplete T-regs and subsequently enhance the immune reconstitution and reverse post transplant lymphopenia. This may indirectly enhance the efficacy of autologous transplantation and reduce disease relapse.

ELIGIBILITY:
Inclusion Criteria:

All patients age > =18 who have been diagnosed with Multiple Myeloma and are scheduled for autologous peripheral blood hematopoietic stem cell transplant (AHSCT) will be screened for eligibility.

Patients must fulfill all of the following inclusion criteria to be eligible for this study:

1. Diagnosis of Multiple Myeloma
2. Age >=18 and no more than 70 years.
3. Able to understand and sign a consent form.
4. Can collect peripheral blood stem cells with a CD34+ cell dose of at least 5.0 x 106/kg. The CD34 molecule is a Cluster of Differentiation molecule present on hematopoietic stem cells.
5. Conditioning regimen to be high dose Melphalan at a dose of 200mg/m2.
6. Karnofsky Performance Score (KPS) >60 or ECOG (Eastern Cooperative Oncology Group) performance status <=2
7. Kidney function:Creatinine <2.0 mg/dl or creatinine clearance >50 ml/min
8. Heart function: Ejection fraction >45%
9. Liver function tests :Serum bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST) less than 3 X upper limit of normal
10. Lung function tests: Forced Vital Capacity (FVC), Forced Expiratory Volume in One Second (FEV1) or Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) >45% predicted

Exclusion Criteria:

1. Age <18 years or > 70 years
2. Previous exposure to denileukin diftitox.
3. Patients with documented uncontrolled central nervous system (CNS) disease.
4. Previous AHSCT.
5. Significant organ dysfunction deemed to be inappropriate for autologous transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al-Kadhimi, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer center clinic.
Groups:
- Denileukin Diftitox (Ontak): Denileukin Diftitox (Ontak) administered Post Autologous Transplantation.
  Denileukin Diftitox (Ontak) : After receiving their stem cell transplant on Day 0, participants will receive study agent via a 30 minute infusion. Participants will also receive a 30 minute infusion of study agent on Day 21.
  Follow-up visits for clinical assessment, blood draws for routine clinical laboratory studies and for immuno-correlative studies will also take place on days 42, 90, 180 and 360.
Period: Overall Study
Arm/Group | Denileukin Diftitox (Ontak)
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Denileukin Diftitox (Ontak)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Assess Toxicities of Giving Two Doses of Ontak at Days 0 and 21 Post Autologous Stem Cell Transplantation in a Dose Escalation Fashion.
Description: After drug infusion, participants will be closely monitored for at least 4 hours for side effects
Time Frame: Up to 21 days post transplant
Arm/Group | Denileukin Diftitox (Ontak)
Number analyzed (Participants) | 0

2. Secondary Outcome: To Evaluate the Effect of Ontak on the Number and Percentage of Regulatory T Cells in the Peripheral Blood Post Transplant at Each Dose Level.
Time Frame: days 0 and 21 post autologous stem cell transplantation
Reporting Status: Not Posted

3. Secondary Outcome: To Evaluate the Effect of Ontak on T Cell CD4/CD8 Reconstitution Post Transplant at Each Dose.
Time Frame: days 0 and 21 post autologous stem cell transplantation
Reporting Status: Not Posted

4. Secondary Outcome: To Evaluate the Effect of Ontak on Engraftment of Neutrophils and Platelets Post Transplant at Each Dose.
Description: During hospitalization stay (approximately 2 weeks), participants will receive injections of G-CSF on a daily basis starting on Day 6 and ending when white blood cells have engrafted. Participants usually remain hospitalized until engraftment.
Time Frame: days 0 and 21 post autologous stem cell transplantation
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Denileukin Diftitox (Ontak)
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denileukin Diftitox (Ontak) (N=2)
Low BUN (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Streptococcus in urine (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Analysis was not completed due to the small number of patients accrued and drugs were unavailable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes